CLINICAL TRIAL: NCT03698448
Title: A Randomized, Double Blind, Dose-finding Study of Inhaled Oligosaccharide (OligoG) vs Placebo in Patients With Cystic Fibrosis
Brief Title: A Dose-finding Study of Inhaled OligoG vs Placebo in Patients With Cystic Fibrosis
Acronym: SMR3372
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Determined not feasible
Sponsor: AlgiPharma AS (Industry)
Collaborators: Imperial College London (Other); Cystic Fibrosis Foundation (Other); European Cystic Fibrosis Society (Unknown); University Hospital of Cologne (Other); Cystic Fibrosis Europe (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3372; 2018-000378-30 (EudraCT Number)
Record Dates: First submitted 2018-10-03; First posted 2018-10-09 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Cystic Fibrosis
Keywords: Oligosaccharide
MeSH Terms: conditions — Cystic Fibrosis | interventions — Inhalation

STUDY DESIGN:
Intervention Model Description: Randomised, double blind, dose-finding
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo medication with identical appearance to the active drug
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo DPI (Placebo Comparator): Matching placebo dry powder for inhalation. OligoG is replaced by lactose. 10 capsules, BID
  Interventions: Drug: OligoG Dry powder for inhalation
- Low dose OligoG DPI (Active Comparator): 17.5 mg OligoG dry powder for inhalation. 10 capsules, BID
  Interventions: Drug: OligoG Dry powder for inhalation
- medium dose OligoG DPI (Active Comparator): 27.5 mg OligoG dry powder for inhalation. 10 capsules, BID
  Interventions: Drug: OligoG Dry powder for inhalation
- High dose OligoG DPI (Active Comparator): 37.5 mg OligoG dry powder for inhalation. 10 capsules, BID
  Interventions: Drug: OligoG Dry powder for inhalation

INTERVENTIONS:
Drug: OligoG Dry powder for inhalation — 10 capsules Dry Powder for Inhalation, BID
  Other Names: Placebo dry powder for inhalation

SUMMARY:
Randomized, double blind, placebo controlled study. The study has two parts:

Dose-finding part, followed by longer term follow-up (6 months)

DETAILED DESCRIPTION:
Part 1: Randomized, double blind, placebo controlled dose-finding. Patients will be assigned to 1 of 3 doses OligoG, or to placebo, on top of Standard of Care. Patients will be treated for 12 weeks, followed by 4 weeks washout.The primary endpoint is relative change in % predicted FEV1. Secondary endpoints include additional spirometry parameters, exacerbation rate, Quality of Life, sputum rheology and microbiology, safety laboratory tests and adverse event reporting.

Part 2: Randomized double-blind 6 -month study, for longer term follow-up of the dose identified in Part 1. New patients will be recruited in part 2, in addition to patients who received placebo in Part 1. In addition to the endpoints studied in Part 1, Part 2 will include Lung Clearance Index (LCI), chest imaging by MRI or CT, and pharmaco-economic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF
* FEV1 at screening >40 and < 90% of predicted normal
* History of PA infection in last 12 m
* History of antibiotic treatment due tp PA infection (not for eradication) during last 12 m
* Concomitant inhaled tobramycin, colistin, aztreonam, or levoflaxin (cycled or continuous)
* Stable CF disease
* Willing to remain on stable CF medication (Standard of care)
* Women of child-bearing potential must habe negative urine pregnany test
* Males & females must use acceptable contraception
* Capable of inhaling dry powder
* willing to sign informed consent
* willing and able to follow study procedures

Exclusion Criteria:

* Use of hypertonic saline > twice daily
* Clinically significant abnormal lab findings, except CRP. In case of high GGT values, case will be discussed by experts before deciding
* History of comorbidity that may distort results or cause additional risk
* pulmonary exacerbation within 28 days prior to randomisation
* Change in CF therapy within 28 days prior to randomisation
* Burkholderia spp. finding within 12 m prior to screening
* pregnant or breast feeding females
* History of allergic reactions to IMP ingredients, incl milk protein
* Inability to perform lung function tests according to ATS/ ERS criteria
* Uncontrolled or unstable diseases that might limit compliance
* History of, or planned organ transplantation
* Allergic ABPA in the last 12 months prior to the screening visit
* Requirement for continuous oxygen supplementation
* Current participation in another clinical study
* medical condition, other than CFwhich exposes the patient to an unacceptably high risk
* Concurrent mlignant disease, except BCC and cervical neoplasia
* Clinically significant alcohol or drug abuse

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) | Change from before to after 12 weeks treatment (Part 1) and 26 weeks (Part 2)
  the amount of air a person can forcefully exhale in one second

SECONDARY OUTCOMES:
Lung Clearance Index (LCI) (Part two only) | Change from before to after 26 weeks treatment
  Lung clearance index (LCI) measured by multiple breath washout is a sensitive measure of ventilation inhomogeneity.
Sputum culture microbiology | Change from before to after 12 weeks treatment (Part 1) and 26 weeks (Part 2)
  Reduction in Pseudomonas Aeruginosa CFU Counts and total counts
Pulmonary Exacerbations | Change from before to after 12 weeks treatment (Part 1) and 26 weeks (Part 2)
  Acute pulmonary exacerbations

CONTACTS AND LOCATIONS:
Overall Officials: Silke van Koningsbruggen-Rietschel, MD, PhD, Principal Investigator — University Hospital Cologne
Locations (1):
- CF Zentrum Köln, Universitätskrankenhaus Köln, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No